CLINICAL TRIAL: NCT02072421
Title: A Prospective, Multi-center, Non-Randomized, Single-arm, Open-label Study of Percutaneous Coronary Intervention in Community Hospitals Without Cardiac Surgery-On-Site
Brief Title: The MASS COMM Post-Randomization Phase Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baim Institute for Clinical Research (Other)
Collaborators: Brockton Hospital (Other); Good Samaritan Hospital Medical Center, New York (Other); Norwood Hospital (Other); Holy Family Hospital, Methuen, MA (Other); Lawrence General Hospital (Unknown); Lowell General Hospital (Other); Melrose Wakefield Hospital (Unknown); Metro West Medical Center (Other); Saints Memorial Medical Center (Unknown); South Shore Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DPH00-Cohort
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-SOS (Other)
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI

SUMMARY:
The primary objective of the Post-Randomization Phase Cohort Study is to continue to assess the safety of non-emergency PCI performed at hospitals without cardiac surgery on-site in patients with myocardial ischemia (other than ST-segment elevation myocardial infarction [STEMI]).

DETAILED DESCRIPTION:
The MASS COMM Post-Randomization Phase Cohort Study ("Cohort Study" is a prospective, multi-center, single-arm study of non-emergency PCI performed at non-SOS hospitals in patients with myocardial ischemia (other than STEMI). The Cohort Study is designed to allow non-SOS hospitals to continue to perform non-emergency PCI after enrollment to the MASS COMM trial is completed and before the 30-day and 12-month results are available.

Specifically, all eligible subjects, after enrollment to the MASS COMM randomized controlled trial is completed and before the final results are available and a decision is reached by the MA-DPH, will be consented and enrolled into this Cohort Study. Subjects will be followed through 30 days post procedure.

ELIGIBILITY:
Inclusion Criteria:

Candidates for this study must meet ALL of the following criteria:

* Subject is at least 18 years old.
* Subject requires single- or multi-vessel percutaneous coronary intervention (PCI) of de novo or restenotic target lesion (including in-stent restenotic lesions). N.B. staged procedure will not be considered to meet the endpoint component of repeat revascularization if either of the following pre-catheterization procedure qualifying clinical laboratory values are met:

  * eGFR is less than 60 ml/min or
  * creatinine is greater than 1.5 mg/dl
* Subject's lesion(s) is (are) amenable to stent treatment with currently available FDA-approved bare metal or drug eluting stents.
* Subject is an acceptable candidate for non-emergency, urgent or emergency CABG.
* Subject has clinical evidence of ischemic heart disease in terms of a positive functional study, or documented symptoms.
* Documented stable angina pectoris [Canadian Cardiovascular Society Classification (CCS) 1, 2, 3, or 4], unstable angina pectoris with documented ischemia (Braunwald Class IB-C, IIB-C, or IIIB-C), non-ST segment elevation myocardial infarction, or documented silent ischemia.
* Subject and the treating physician agree that the subject will comply with all follow-up evaluations.
* Subject has been informed of the nature and purpose of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical site.

Angiographic Inclusion Criteria

* The target lesion(s) is (are) de novo or restenotic (including in-stent restenotic) native coronary artery lesion(s) with greater or equal to 50 and less than 100% stenosis (visual estimate), or the target lesion is an acute (less than 1 month) total occlusion as evidenced by clinical symptoms.
* If Fractional Flow Reserve (FFR) is measured, target lesion(s) has (have) evidence of a hemodynamically significant stenosis determined by FFR measurement (FFR less than or equal to 0.8).
* Target lesions(s) is (are) located in an infarct (if not treated with primary PCI) or non-infarct-related artery with a 70% or greater stenosis (by visual estimate) greater than 72 hours following the STEMI.

Lesions treated with PCI greater than 72 hours following STEMI would be subject to the same protocol inclusion/exclusion criteria listed above and below with the exception that a target lesion of 70% or greater stenosis may be treated with or without symptoms or abnormal stress test).

Exclusion Criteria:

Subjects will be excluded from participation in the Cohort Study (and non-emergency PCI may not be performed in these patients at the non-SOS site) if ANY of the following conditions apply:

* The patient is pregnant or breastfeeding.
* Evidence of ST segment elevation myocardial infarction within 72 hours of the intended treatment on infarct related or non-infarct related artery.
* Cardiogenic shock on presentation or during current hospitalization.
* Left ventricular ejection fraction less than 20%.
* Known allergies to: aspirin, clopidogrel (Plavix), prasugrel (Effient), and ticlopidine (Ticlid), heparin, bivalirudin, stainless steel, or contrast agent (which cannot be adequately premedicated).
* A platelet count less than 75,000 cells/mm3 or greater than 700,000 cells/mm3 or a WBC less than 3,000 cells/mm3.
* Acute or chronic renal dysfunction (creatinine less than 2.5 mg/dl or less than 150µmol/L).
* Subject is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints. (Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials).
* Prior participation in the MASS-COMM Trial, unless the patient has completed the 12-month follow-up for the Trial, and/or prior participation in the Cohort Study, unless the patient has completed the 30-day follow-up for the Cohort Study.
* Within 30 days prior to the index Cohort Study procedure, the subject has undergone a previous coronary interventional procedure of any kind. Note: This exclusion criterion does not apply to post-STEMI patients.
* Stroke or transient ischemic attack within the prior 3 months.
* Active peptic ulcer or upper GI bleeding within the prior 3 months.
* Subject has active sepsis.
* Unprotected left main coronary artery disease (stenosis greater than 50%).
* Subject has evidence of a hemodynamically insignificant stenosis determined by FFR measurement (FFR greater than 0.8).
* In the investigator's opinion, subject has a co-morbid condition(s) that could limit the subject's ability to participate in the study or comply with follow-up requirements or impact the scientific integrity of the study.

Angiographic Exclusion Criteria

* Subject has normal or insignificant coronaries (i.e., coronary lesion(s) less than 50% stenosis).
* Any target vessel has evidence of:

  1. excessive thrombus (e.g., requires target vessel thrombectomy)
  2. tortuosity (greater than 60 degree angle) that makes it unsuitable for proper stent delivery and deployment,
  3. heavy calcification.
* Any target lesion requires treatment with a device other than PTCA prior to stent placement (e.g. but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.).
* Any lesion that is located in a saphenous vein graft, however, lesions located within the native vessel but accessed through the graft are eligible.
* The target vessel is in a "last remaining" epicardial vessel (e.g., >2 non-target epicardial vessels and the bypass grafts to these territories [if present] are totally occluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2879 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice K Jacobs, MD, Principal Investigator — Boston University School of Medicine , Boston Medical Center; Laura Mauri, MD, Principal Investigator — Brigham and Women's Hospital; Sharon-Lise Normand, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (10):
- United States (10):
  - Good Samaritan Medical Center, Brockton, Massachusetts
  - Brockton Hospital, Brockton, Massachusetts
  - Metrowest Medical Center, Framingham, Massachusetts
  - Lawrence General Hospital, Lawrence, Massachusetts
  - Saints Memorial Medical Center, Lowell, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Melrose-Wakefield Hospital, Melrose, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Norwood Hospital, Norwood, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- PCI at Hospitals Without On-Site Cardiac Surgery: PCI at a hospital without on-site cardiac surgery
Period: Overall Study
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery
Started | 2879
Completed | 2489
Not Completed | 390

BASELINE CHARACTERISTICS:
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery
Number analyzed (Participants) | 2879
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.92 (11.48)
Sex/Gender, Customized [Number; unit: participants]
  Male | 1955
  Female | 924
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 2595
  Black | 61
  Hispanic | 153
  Asian | 50
  Native American | 1
  Other | 19

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiac Event (MACE)
Description: MACE is a composite of all cause mortality, myocardial infarction (Q wave and non-Q wave), repeat coronary revascularization (of the target vessel or non-target vessel) by either percutaneous or coronary artery bypass graft (CABG) methods, or stroke, at 30-days.
Time Frame: 30-days
Measure: Number; unit: participants
Groups:
- PCI at Hospitals Without On-Site Cardiac Surgery: Assigned to PCI at a hospital without on-site cardiac surgery
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery
Number analyzed (Participants) | 2879
participants | 229

2. Secondary Outcome: All-Cause Mortality
Description: all-cause mortality through 30 days post-procedure
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery
Number analyzed (Participants) | 2879
participants | 15

3. Secondary Outcome: Stroke
Description: Stroke through 30 days post-procedure
Time Frame: 30 days
Measure: Number; unit: participants
Groups:
- PCI at a Hospital Without On-site Cardiac Surgery: PCI at a hospital without on-site cardiac surgery
Arm/Group | PCI at a Hospital Without On-site Cardiac Surgery
Number analyzed (Participants) | 2879
participants | 2

4. Secondary Outcome: Revascularization
Description: Repeat coronary revascularization including emergency or urgent revascularization through 30 days post-procedure
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | PCI at a Hospital Without On-site Cardiac Surgery
Number analyzed (Participants) | 2879
participants | 75

5. Secondary Outcome: Major Vascular Complications
Description: Major vascular complications, including access site complications and major bleeding events requiring transfusion,through 30 days post-procedure.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | PCI at a Hospital Without On-site Cardiac Surgery
Number analyzed (Participants) | 2879
participants | 28

ADVERSE EVENTS:
Description: Serious and other adverse events were not collected in this study.
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No